CLINICAL TRIAL: NCT00681512
Title: Berry Interventional Trial (BIT) in Resected Non-Small Cell Lung Cancer
Brief Title: The Effect of Berries on Lung Cancer Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Ramesh Gupta, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08.0040; BCC-LUN-07-002 (Other: Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; lung cancer; non small cell lung cancer; lung carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: berry powder — All subjects (lung cancer survivors and volunteers) will consume 20 grams of berry powder (blueberries, black raspberries, or a mixture of both) per day by mouth for the first 3 days, then 40 grams of berry powder by mouth every day for 4 to 5 weeks.
  The berry powder is to be mixed in subject's routine intake of milk, yogurt, juice, or water.
  All subjects will have the option to continue the berry regimen for an extended period. Subjects who choose to do so will not consume any berry powder for one week. After one week, subjects will begin consuming 40 grams of the berry powder every day for an additional 4 to 5 weeks.
  Other Names: berries; berry

SUMMARY:
The purpose of this study is to determine how berries affect cancer tumors in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
In the United States, more people (161,840 per year) die of lung cancers than of prostate cancer, breast cancer and colon cancer combined. Presently, there are over 43 million current smokers and over 47 million ex-smokers living in the US. Due to the lag time between smoking and the development of cancer, there are significant numbers of ex-smokers and current smokers who may develop lung cancer compared to never smokers.

Recent studies in animals have shown that berries, given as a dietary supplement, are highly effective against certain types of cancers. In a study involving mice with lung tumors, mice that had consumed a mixture of berries developed fewer tumors and had less tumor growth than mice that did not consume berries.

The berries used in this study will consist of blueberries, black raspberries, or a mixture of both.

ELIGIBILITY:
Inclusion Criteria (lung cancer survivors):

* men treated for lung cancer, women treated for lung cancer and with no child-bearing potential (hysterectomy, tubal ligation, post-menopausal women)

Exclusion Criteria (lung cancer survivors):

* women who are on hormone replacement therapy
* women who are pregnant, or planning for pregnancy
* history of lung transplant
* prison inmate
* inability to take oral medication or food
* known or suspected allergy to berries or berry products
* HIV patients

Inclusion Criteria (volunteers):

* adult men, adult women with no child bearing potential (hysterectomy, tubal ligation, post-menopausal women)

Exclusion Criteria (volunteers):

* women who are on hormone replacement therapy
* women who are pregnant, or planning for pregnancy
* history of lung transplant
* prison inmate
* inability to take oral medication or food
* known or suspected allergy to berries or berry products
* HIV patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assessment of blueberry and black raspberry phenolics in plasma and urine | upon completion of 4 to 5 weeks of daily consumption of berry powder
  In addition to determining the berry phytochemical profile in plasma and urine, this study will attempt to establish the effect of berries on modulating immunological profiles such as the complete blood count, and T, B and natural killer (NK) cell populations and circulating biomarkers (serum proteins and microRNAs). This pilot study will establish the safety and feasibility of conducting a larger clinical trial with berry intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Gupta, PhD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States